CLINICAL TRIAL: NCT01857622
Title: Phase III Clinical Study of DU-176b (Non-valvular Atrial Fibrillation): Japanese, Multicenter, Open-label Study of DU-176b in Patients With Non-valvular Atrial Fibrillation and Severe Renal Impairment (SRI)
Brief Title: Safety and Pharmacokinetics Study of DU-176b Administered to Non-valvular Atrial Fibrillation With Severe Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DU176b-B-J307
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2015-01

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: anticoagulant; DU-176b; edoxaban; factor Xa; oral; atrial fibrillation; severe renal impairment
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SRI 15mg (Experimental): DU-176b was orally administered at a dose of 15 mg once daily for 12 weeks.
  Interventions: Drug: DU-176b 15mg
- Normal/MiRI low-dose group (Experimental): DU-176b was orally administered at a dose of 30 mg once daily for 12 weeks in subjects who had none of the dose adjustment factors (body weight of ≤ 60 kg or the presence of concurrent treatment with quinidine or verapamil). DU-176b was orally administered at a dose of 15 mg once daily for 12 weeks to subjects who had any of the dose adjustment factors, irrespective of the number of dose adjustment factors.
  Interventions: Drug: DU-176b 30mg
- Normal/MiRI high-dose group (Experimental): DU-176b was orally administered at a dose of 60 mg once daily for 12 weeks in subjects who had none of the dose adjustment factors. DU-176b was orally administered at a dose of 30 mg once daily for 12 weeks to subjects who had any of the dose adjustment factors, irrespective of the number of dose adjustment factors.
  Interventions: Drug: DU-176b 60mg

INTERVENTIONS:
Drug: DU-176b 15mg — oral DU-176b 15mg once daily
  Other Names: edoxaban
  Arms: SRI 15mg
Drug: DU-176b 30mg — oral DU-176b 30mg once daily
  Other Names: edoxaban
  Arms: Normal/MiRI low-dose group
Drug: DU-176b 60mg — oral DU-176b 60mg once daily
  Other Names: edoxaban
  Arms: Normal/MiRI high-dose group

SUMMARY:
To assess the safety and pharmacokinetics of DU-176b administered to non-valvular atrial fibrillation patients with severe renal impairment, compared with DU-176b administered to non-valvular atrial fibrillation (NVAF) patients with normal renal function or mild renal impairment (Normal/MiRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with NVAF and SRI, or patients with NVAF and Normal/MiRI.

Exclusion Criteria:

* Patients who are on hemodialysis or patients who may start hemodialysis before the follow-up assessment
* Patients who are at a significantly high risk for bleeding
* Patients who are receiving treatment with any anticoagulant drugs excluding warfarin, rivaroxaban, and dabigatran
* Patients who have evidence of hepatic function test abnormalities

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yukihiro Koretsune, Dir, Principal Investigator — Osaka National Hospital
Locations (1):
- Tokyo Women's Medical University Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Groups:
- SRI 15mg: Severe Renal Impairment DU-176b was orally administered at a dose of 15 mg once daily for 12 weeks.
  DU-176b 15mg: oral DU-176b 15mg once daily
- Normal/MiRI Low-dose Group: Normal or Mild Renal impairment DU-176b was orally administered at a dose of 30 mg once daily for 12 weeks in subjects who had none of the dose adjustment factors (body weight of ≤ 60 kg or the presence of concurrent treatment with quinidine or verapamil). DU-176b was orally administered at a dose of 15 mg once daily for 12 weeks to subjects who had any of the dose adjustment factors, irrespective of the number of dose adjustment factors.
  DU-176b 30mg: oral DU-176b 30mg once daily
- Normal/MiRI High-dose Group: Normal or Mild Renal Impairment DU-176b was orally administered at a dose of 60 mg once daily for 12 weeks in subjects who had none of the dose adjustment factors. DU-176b was orally administered at a dose of 30 mg once daily for 12 weeks to subjects who had any of the dose adjustment factors, irrespective of the number of dose adjustment factors.
  DU-176b 60mg: oral DU-176b 60mg once daily
Period: Overall Study
Arm/Group | SRI 15mg | Normal/MiRI Low-dose Group | Normal/MiRI High-dose Group
Started | 50 | 22 | 21
Completed | 39 | 21 | 19
Not Completed | 11 | 1 | 2
Not completed — Adverse Event | 5 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 4 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SRI 15mg | Normal/MiRI Low-dose Group | Normal/MiRI High-dose Group | Total
Number analyzed (Participants) | 50 | 22 | 21 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.9 (6.04) | 68.0 (8.91) | 72.2 (4.58) | 75.9 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 4 | 7 | 33
  Male | 28 | 18 | 14 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 50 | 22 | 21 | 93
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 50 | 22 | 21 | 93

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Any Adjudicated Bleeding Events
Description: Incidence of any adjudicated bleeding events (including major bleeding, clinically relevant non-major bleeding, and minor bleeding)
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleeds
Arm/Group | SRI 15mg | Normal/MiRI Low-dose Group | Normal/MiRI High-dose Group
Number analyzed (Participants) | 50 | 22 | 21
percentage of subjects with bleeds | 20.0 [11.2 to 33.0] | 22.7 [10.1 to 43.4] | 23.8 [10.6 to 45.1]
Statistical Analysis 1: Comparison: SRI 15mg vs Normal/MiRI High-dose Group; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); no statistical test; Cox Proportional Hazard = 3.8, 95% CI 2-sided [-14.7 to 26.8]
Statistical Analysis 2: Comparison: SRI 15mg vs Normal/MiRI Low-dose Group; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Cox Proportional Hazard = 2.7, 95% CI 2-sided [-15.4 to 25.2]

ADVERSE EVENTS:
Arm/Group | SRI 15mg | Normal/MiRI Low-dose Group | Normal/MiRI High-dose Group
Serious Adverse Events (participants affected / at risk) | 5/50 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 33/50 | 14/22 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SRI 15mg (N=50) | Normal/MiRI Low-dose Group (N=22) | Normal/MiRI High-dose Group (N=21)
pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SRI 15mg (N=50) | Normal/MiRI Low-dose Group (N=22) | Normal/MiRI High-dose Group (N=21)
nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4) | 5 (5)
pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
gingival bleeding (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0)
haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 4 (4)
Blood creatinine increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
occult blood (Investigations) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetit (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the results of the Study at any time without the prior written approval of Sponsor.